CLINICAL TRIAL: NCT05561881
Title: Comparison of Efficacy Between Ultra-sound Genicular Nerve Block Versus the Popliteal Artery and the Capsule of the Posterior Knee(IPACK) Block for Knee Arthroscopic Surgery
Brief Title: Genicular Nerve Block Versus IPACK Block for Knee Arthroscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amani Hassan Abdel-Wahab, assistant professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AssiutU_HA
Record Dates: First submitted 2022-09-28; First posted 2022-09-30 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Genicular Nerve Block
MeSH Terms: interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IPACK group (Other): visualization of the popliteal artery and posterior surface of the distal femur then the image of the femoral condyles and popliteal artery will be obtained. A needle with a tip length of 100 mm will be inserted in a medial to a lateral plane parallel to the femur in the middle area between the popliteal artery and femur,20 ml local anesthetic solution will be given into this space with adequate and equal distribution of anesthetic agent
  Interventions: Other: popliteal artery and the capsule of the posterior knee (IPACK) block
- genicular group (Experimental): US transducer placed parallel to the femur shaft and the epicondyle will be identified, the superomedial superolateral and inferomedial genicular arteries, which follow a similar route with each genicular nerve will be visualized close to the periosteal areas, and A 20G needle with a tip length of 50mm will be directed in the plane of the US probe in the long axis view. After confirming the placing of the needle next to each genicular artery a total amount of 20 ml of local anesthetic in equal increments at multiple sites
  Interventions: Other: genicular nerves block

INTERVENTIONS:
Other: popliteal artery and the capsule of the posterior knee (IPACK) block — ultra-sound visualization of the popliteal artery and posterior surface of the distal femur then the image of the femoral condyles and popliteal artery will be obtained. A needle with a tip length of 100 mm will be inserted in a medial to the lateral plane parallel to the femur in the middle area between the popliteal artery and femur,20 ml local anesthetic solution will be given into this space with adequate and equal distribution of anesthetic agent
  Arms: IPACK group
Other: genicular nerves block — ultra-sound transducer placed parallel to the femur shaft and the epicondyle will be identified, the superomedial superolateral and inferomedial genicular arteries, which follow a similar route with each genicular nerve will be visualized close to the periosteal areas, A20G needle with a tip length of 50mm will be directed in the plane of the US probe in the long axis view. After confirming placing of the needle next to each genicular artery a total amount of 20 ml local anesthetic in equal increments at multiple sites.
  Arms: genicular group

SUMMARY:
Postoperative pain management after knee arthroscopic surgery continues to evolve with better treatment strategies being formulated to improve patient satisfaction, and clinical outcomes and reduce opioid use in the immediate postoperative period. appropriate perioperative pain management has been shown to result in faster recovery and rehabilitation leading to better functional outcomes in patients undergoing knee arthroscopic surgery. this has necessitated the development of multimodal analgesics. peripheral nerve blockade has been reported to deliver optimal postoperative pain relief and is increasingly preferred in patients undergoing arthroscopic procedures and various different techniques such as sciatic nerve block, femoral nerve block, and genicular block have been described.

DETAILED DESCRIPTION:
The genicular nerves include branches from the femoral, common peroneal, saphenous, tibial, and obturator nerves which innervate the knee capsule. the superolateral, superomedial, and inferomedial branches of the genicular nerve were reported to be in proximity to the periosteum of the tibia and femur, and the superolateral, inferolateral, superomedial, and inferomedial quadrant of the anterior knee joint were shown to be innervated by superior lateral, inferior lateral, superior medial and inferior medial branches of the genicular nerve, respectively alongside the branches of peroneal and femoral nerves Thus, a genicular nerve block specifically Targets these branches which innervate the knee joint for the management of postoperative pain in arthroscopic surgery.

On the other hand, the interspace between the popliteal artery and capsule of the knee(IPACK) block provides analgesia on the posterior knee joint, and the application of a genicular or IPACK block has been proven to be associated with promising outcomes following arthroscopic surgery

ELIGIBILITY:
Inclusion Criteria:

* age 20_60 years
* American Society of anthologist class I-III
* BMI18_35 kg/m2
* scheduled for primary unilateral knee arthroscopic surgery

Exclusion Criteria:

* known allergy to local anesthesia
* contraindication to local anesthesia injection (e.g., infection at the site of injection
* contraindication to spinal anesthesia (e.g., coagulopathy)
* patients with preexisting motor or sensory deficit in lower extremities
* insulin or non-insulin-dependent diabetes mellitus
* systemic corticosteroids use within 30 days
* history of arrhythmia or seizures
* severe renal insufficiency
* patient refusal

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Pain Visual Analogue Scale (VAS) | first postoperative 24 hours
  VAS in the first postoperative 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Amani H Abdel-wahab, MD, Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No